CLINICAL TRIAL: NCT00745615
Title: An Active Extension of LAQ/5062 Study. A Multinational, Multicenter, Randomized, Double-Blind, Parallel-Group Study to Evaluate the Safety, Tolerability and Efficacy of Two Doses (0.3 mg and 0.6 mg) of Laquinimod, Orally Administered in Relapsing Remitting (R-R) Multiple Sclerosis (MS) Subjects (Study LAQ/5063 Active Double-Blind Phase) Followed by an Open Label Phase of Laquinimod 0.6 mg Daily (LAQ/5063 OL)
Brief Title: An Extension Study of LAQ/5062 Exploring the Long Term Safety, Tolerability and Clinical Effect Parameters During the Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated RRMS studies as sufficient long term clinical data was collected for the study drug in the relevant dose.
Sponsor: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAQ/5063OL; LAQ/5063 (Other: Sponsor ID); 2005-004334-41 (EudraCT Number)
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding performed by interactive voice response system (IVRS) and relevant only to the first period of the extension. General medical evaluations will be assessed separately from neurological assessment evaluations by two different neurologists/ physicians. Magnetic resonance imaging (MRI) scan evaluation will be performed at a central reading center by staff that does not have access to the clinical data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Double-Blind: Laquinimod 0.3 mg (Experimental): Participants who will be receiving laquinimod 0.3 milligram (mg) tablet once daily orally in double-blind core study, will continue to receive laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
  Interventions: Drug: Laquinimod
- Double-Blind: Laquinimod 0.6 mg (Experimental): Participants who will be receiving laquinimod 0.6 mg (2 tablets of 0.3 mg each) once daily orally in double-blind core study, will continue to receive laquinimod 0.6 mg once daily orally in double-blind extension period of this study for up to Week 36.
  Interventions: Drug: Laquinimod
- Double-Blind: Placebo/Laquinimod 0.3 mg (Experimental): Participants who will be receiving placebo matching to laquinimod 0.3 mg tablet once daily orally in double-blind core study, will receive laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Double-Blind: Placebo/Laquinimod 0.6 mg (Experimental): Participants who will be receiving placebo matching to laquinimod 0.6 mg (2 tablets of placebo) once daily orally in double-blind core study, will receive laquinimod 0.6 mg once daily orally in double-blind extension period of this study for up to Week 36.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg (Experimental): Participants who will be receiving laquinimod 0.3 mg tablet once daily orally either in double-blind core study or double-blind extension period, will receive laquinimod 0.6 mg capsule once daily orally in open-label extension period of this study until termination (as long as the Sponsor will continue the development of laquinimod 0.6 mg for RRMS) or early discontinuation (up to approximately 10.5 years).
  Interventions: Drug: Laquinimod
- Open Label: Laquinimod 0.6 mg (Experimental): Participants who will be receiving laquinimod 0.6 mg (2 tablets of 0.3 mg each) once daily orally either in double-blind core study or double-blind extension period, will receive laquinimod 0.6 mg capsule once daily orally in open-label extension period of this study until termination (as long as the Sponsor will continue the development of laquinimod 0.6 mg for RRMS) or early discontinuation (up to approximately 10.5 years).
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Laquinimod — Laquinimod tablets/capsules will be administered as per the dose and schedule specified in the respective arms.
  Other Names: TV-5600
Drug: Placebo — Placebo matching to laquinimod will be administered as per the dose and schedule specified in the respective arms.
  Arms: Double-Blind: Placebo/Laquinimod 0.3 mg; Double-Blind: Placebo/Laquinimod 0.6 mg

SUMMARY:
This is a multinational, multicenter, randomized, double-blind, parallel-group active extension of LAQ/5062 study (NCT00349193), assessing the tolerability, safety and efficacy of two doses (0.3 mg and 0.6 mg) of laquinimod, orally administered in participants with relapsing remitting multiple sclerosis (RRMS), followed by an open-label phase of laquinimod 0.6 mg daily. This study is LAQ/5063 (i.e., double-blind extension) and LAQ/5063 OL (i.e., subsequent open-label extension). - The first period of the extension study is an active, double-blind period. Participants from the active treatment arms in LAQ/5062 continue their assigned treatment in blinded fashion. Participants who were assigned to placebo treatment in LAQ/5062 are equally randomized in blinded-fashion to laquinimod 0.6 mg or laquinimod 0.3 mg. - Once termination visit of LAQ/5063 active double-blind phase (completion of the full 36 weeks or as requested by the Sponsor) is performed, all participants continue on laquinimod 0.6 mg daily as an open-label intervention. The open-label period continues as long as the Sponsor continues the development of laquinimod 0.6 mg for RRMS or early discontinuation.

ELIGIBILITY:
Inclusion Criteria - Participants must have completed the 36 weeks of treatment (completion of the full 36 weeks or as requested by the Sponsor) of the active double-blind phase. - Women of childbearing potential (for example, women who were not postmenopausal or surgically sterilized) must have practiced 2 acceptable methods of birth control for the duration of the study and until 30 days after the last dose of study medication (acceptable methods of birth control in this open-label extension phase included intrauterine devices, barrier methods [condom or diaphragm with spermicide], and hormonal methods of birth control [for example, oral contraceptive, contraceptive patch, and long-acting injectable contraceptive]). - Participants must have been willing and able to comply with the protocol requirements for the duration of LAQ/5063 OL. - Participants must have given signed, written informed consent prior to entering LAQ/5063 OL. - For the 36 months further extension: Participants must have completed the 24 months of treatment of the first period of the open label phase. Exclusion Criteria - For the 36 month further extension: Premature discontinuation from LAQ/5063 OL phase prior to completion of 24 months of treatment period. - Pregnancy or breastfeeding. - Participants with clinically significant or unstable medical or surgical condition, detected or worsened during the active double-blind phase of LAQ/5063, which would have precluded safe and complete study participation. - Use of experimental drugs, immunosuppressive drugs, and/or participation in clinical studies within the period from termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Previous treatment with immunomodulators with the exception of laquinimod (including interferon [IFN] 1a and 1b, glatiramer acetate, and intravenous [IV] immunoglobulin) within 2 months prior to entering the open-label phase for those subjects who had a time gap between termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Use of corticosteroids within 30 days prior to entering the open-label phase, except for IV methylprednisolone 1 grams/day for a maximum of 3 days, in the period from termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Use of potent inhibitors of cytochrome P3A4 (CYP3A4) within 2 weeks prior to LAQ/5063 OL and/or use of fluoxetine 1 month prior to entering LAQ/5063 OL, in the period from termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Use of the following substrates of cytochrome P1A2 (CYP1A2): theophylline and/or warfarin within 2 weeks prior to entering LAQ/5063 OL, in the period from termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Use of amiodarone in the period from termination of LAQ/5063 active double-blind phase to LAQ/5063 OL. - Following the switch to new formulation (capsules), hypersensitivity to mannitol, meglumine, or sodium stearyl fumarate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2005-12-07 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, Principal Investigator — Instituto Scientifico Fondazione Centro S. Raffaele, Milan, Italy
Locations (45):
- Czechia (3):
  - Teva Investigational Site 382, Hradec Králové
  - Teva Investigational Site 380, Prague
  - Teva Investigational Site 384, Praha 5- Motol
- Germany (6):
  - Teva Investigational Site 681, Berlin
  - Teva Investigational Site 684, Erfurt
  - Teva Investigational Site 687, Hamburg
  - Teva Investigational Site 683, Mainz
  - Teva Investigational Site 686, Ulm
  - Teva Investigational Site 685, Würzburg
- Hungary (4):
  - Teva Investigational Site 580, Debrecen
  - Teva Investigational Site 581, Gyula
  - Teva Investigational Site 583, Miskolc
  - Teva Investigational Site 584, Veszprém
- Israel (3):
  - Teva Investigational Site 981, Ramat Gan, IL
  - Teva Investigational Site 982, Haifa
  - Teva Investigational Site 980, Jerusalem
- Italy (4):
  - Teva Investigational Site 483, Cagliari
  - Teva Investigational Site 484, Milan
  - Teva Investigational Site 486, Milan
  - Teva Investigational Site 488, Siena
- Poland (6):
  - Teva Investigational Site 281, Bydgoszcz
  - Teva Investigational Site 280, Katowice
  - Teva Investigational Site 285, Katowice
  - Teva Investigational Site 283, Lodz
  - Teva Investigational Site 284, Lublin
  - Teva Investigational Site 282, Wroclaw
- Russia (9):
  - Teva Investigational Site 186, Moscow
  - Teva Investigational Site 187, Moscow
  - Teva Investigational Site 188, Moscow
  - Teva Investigational Site 189, Moscow
  - Teva Investigational Site 180, Saint Petersburg
  - Teva Investigational Site 181, Saint Petersburg
  - Teva Investigational Site 182, Saint Petersburg
  - Teva Investigational Site 184, Saint Petersburg
  - Teva Investigational Site 185, Saint Petersburg
- Spain (6):
  - Teva Investigational Site 782, Barakaldo
  - Teva Investigational Site 785, Barcelona
  - Teva Investigational Site 781, Bilbao
  - Teva Investigational Site 784, L'Hospitalet de Llobregat
  - Teva Investigational Site 780, Madrid
  - Teva Investigational Site 783, Seville
- United Kingdom (4):
  - Teva Investigational Site 884, Liverpool
  - Teva Investigational Site 882, London
  - Teva Investigational Site 881, Sheffield
  - Teva Investigational Site 883, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is LAQ/5063 (i.e., double-blind extension) and LAQ/5063OL (i.e., subsequent open-label extension). Participants who completed double-blind core study LAQ/5062 (NCT00349193) and agreed to continue in active extension study were enrolled in this study.
Pre-assignment Details: Double-blind extension: Participants treated with placebo in LAQ/5062 study were equally randomized to one of 2 groups: Laquinimod 0.6 mg or Laquinimod 0.3 mg. Participants previously treated with laquinimod 0.6 mg or laquinimod 0.3 mg continued on their original treatment. Open-label extension: All participants received laquinimod 0.6 mg.
Groups:
- Double-Blind: Laquinimod 0.3 mg: Participants who were receiving laquinimod 0.3 milligram (mg) tablet once daily orally in double-blind core study, were continued to receive laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
- Double-Blind: Laquinimod 0.6 mg: Participants who were receiving laquinimod 0.6 mg (2 tablets of 0.3 mg each) once daily orally in double-blind core study, were continued to receive laquinimod 0.6 mg once daily orally in double-blind extension period of this study for up to Week 36.
- Double-Blind: Placebo/Laquinimod 0.3 mg: Participants who were receiving placebo matched to laquinimod 0.3 mg tablet once daily orally in double-blind core study, received laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
- Double-Blind: Placebo/Laquinimod 0.6 mg: Participants who were receiving placebo matched to laquinimod 0.6 mg (2 tablets of placebo) once daily orally in double-blind core study, received laquinimod 0.6 mg once daily orally in double-blind extension period of this study for up to Week 36.
- Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg: Participants who were receiving laquinimod 0.3 mg tablet once daily orally either in double-blind core study or double-blind extension period, received laquinimod 0.6 mg capsule once daily orally in open-label extension period of this study until termination (as long as the Sponsor continued the development of laquinimod 0.6 mg for relapsing-remitting multiple sclerosis [RRMS]) or early discontinuation (up to approximately 10.5 years).
- Open Label: Laquinimod 0.6 mg: Participants who were receiving laquinimod 0.6 mg (2 tablets of 0.3 mg each) once daily orally either in double-blind core study or double-blind extension period, received laquinimod 0.6 mg capsule once daily orally in open-label extension period of this study until termination (as long as the Sponsor continued the development of laquinimod 0.6 mg for RRMS) or early discontinuation (up to approximately 10.5 years).
Period: Double-Blind Extension (36 Weeks)
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg | Open Label: Laquinimod 0.6 mg
Started | 80 | 94 | 39 | 44 | 0 | 0
Completed | 75 | 87 | 38 | 39 | 0 | 0
Not Completed | 5 | 7 | 1 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 1 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Than Specified | 0 | 1 | 0 | 0 | 0 | 0
Period: Open-Label (up to Approx 10.5 Years)
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg | Open Label: Laquinimod 0.6 mg
Started | 0 | 0 | 0 | 0 | 96 | 113
Completed | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 91 | 108
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 50 | 50
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 19 | 19
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 9 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 8
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 8 | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who entered in extension study LAQ/5063 (after completion of the entire treatment period in LAQ/5062) and received at least one dose of laquinimod (either 0.3 mg or 0.6 mg) during the active double-blind phase.
Groups:
- Double-Blind: Laquinimod 0.3 mg: Participants who were receiving laquinimod 0.3 mg tablet once daily orally in double-blind core study, were continued to receive laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
- Total: Total of all reporting groups
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg | Total
Number analyzed (Participants) | 80 | 94 | 39 | 44 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (8.3) | 33.4 (8.7) | 34.5 (8.8) | 31.0 (6.6) | 33.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 23 | 27 | 154
  Male | 29 | 41 | 16 | 17 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 1 | 0 | 0 | 0 | 1
  Black of African Heritage | 0 | 1 | 0 | 0 | 1
  Caucasian | 79 | 93 | 39 | 44 | 255
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 8 | 7 | 3 | 3 | 21
  Germany | 7 | 7 | 5 | 3 | 22
  Hungary | 7 | 7 | 3 | 3 | 20
  Israel | 3 | 3 | 3 | 2 | 11
  Italy | 8 | 9 | 2 | 4 | 23
  Poland | 19 | 21 | 11 | 9 | 60
  Russia | 18 | 28 | 9 | 14 | 69
  Spain | 7 | 8 | 3 | 5 | 23
  United Kingdom | 3 | 4 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Extension Period: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline (Week 0) to Week 36
Population: ITT analysis set included all participants who entered in extension study LAQ/5063 (after completion of the entire treatment period in LAQ/5062) and received at least one dose of laquinimod (either 0.3 mg or 0.6 mg) during the active double-blind phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 80 | 94 | 39 | 44
Participants | 57 | 66 | 23 | 32

2. Primary Outcome: Open-label Extension Period: Number of Participants With AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline (Month 0/termination visit of double-blind extension phase [completion of full 36 weeks] until termination (as long as the Sponsor continued the development of laquinimod 0.6 mg for RRMS) or early discontinuation (up to approximately 10.5 years)
Population: Safety analysis set included all participants who had received at least 1 dose of study drug during the open-label extension period LAQ/5063OL.
Measure: Count of Participants; unit: Participants
Groups:
- Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg: Participants who were receiving laquinimod 0.3 mg tablet once daily orally either in double-blind core study or double-blind extension period, received laquinimod 0.6 mg capsule once daily orally in open-label extension period of this study until termination (as long as the Sponsor continued the development of laquinimod 0.6 mg for RRMS) or early discontinuation (up to approximately 10.5 years).
Arm/Group | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg | Open Label: Laquinimod 0.6 mg
Number analyzed (Participants) | 96 | 113
Participants | 86 | 100

3. Primary Outcome: Double-Blind Period: Number of Participants Who Prematurely Discontinued From the Study Due to Any Reason and Due to AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline (Week 0) to Week 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 80 | 94 | 39 | 44
Participants
  Due to any reason | 5 | 7 | 1 | 5
  Due to AEs | 2 | 3 | 1 | 1

4. Primary Outcome: Open-Label Period: Number of Participants Who Prematurely Discontinued From the Study Due to Any Reason and Due to AEs
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg | Open Label: Laquinimod 0.6 mg
Number analyzed (Participants) | 96 | 113
Participants
  Due to any reason | 91 | 108
  Due to AEs | 1 | 9

5. Secondary Outcome: Double-Blind Period: Relapse Rate: Total Number of Confirmed Relapses
Description: Relapse was defined as the appearance of one or more new neurological abnormalities or the reappearance of one or more previously observed neurological abnormalities, lasting for at least 48 hours (in the absence of fever or any infection) and immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. An event was counted as a relapse only when the participant's symptoms were accompanied by observed objective neurological changes, consistent with an increase of at least 0.5 in the Expanded disability status scale (EDSS); or one grade in the score of 2 or more of the 7 Functional Systems (FS) (excluding changes in bowel or bladder function or cognition); or 2 grades in the score of one of the FS as compared to the previous evaluation. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]).
Time Frame: Baseline (Week 0) up to end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 80 | 94 | 39 | 44
relapses | 0.39 (0.68) | 0.36 (0.58) | 0.38 (0.54) | 0.39 (0.72)

6. Secondary Outcome: Double-Blind Period: Percentage of Relapse-Free Participants
Description: Relapse was defined as the appearance of one or more new neurological abnormalities or the reappearance of one or more previously observed neurological abnormalities, lasting for at least 48 hours (in the absence of fever or any infection) and immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. An event was counted as a relapse only when the participant's symptoms were accompanied by observed objective neurological changes, consistent with an increase of at least 0.5 in the EDSS; or one grade in the score of 2 or more of the 7 FS (excluding changes in bowel or bladder function or cognition); or 2 grades in the score of one of the FS as compared to the previous evaluation. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Baseline (Week 0) up to end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 80 | 94 | 39 | 44
percentage of participants | 70.0 | 68.1 | 64.1 | 72.7

7. Secondary Outcome: Double-Blind Period: Number of Enhancing Lesions on T1-Weighted Images
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of gadolinium-enhanced T1 lesions. T1-weighted scan was taken after administration of gadolinium-gadopentetic acid (Gd-DTPA).
Time Frame: At the end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: ITT analysis set included all participants who entered in extension study LAQ/5063 (after completion of the entire treatment period in LAQ/5062) and received at least one dose of laquinimod (either 0.3 mg or 0.6 mg) during the active double-blind phase. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 66 | 82 | 36 | 38
lesions | 2.50 (4.77) | 2.18 (5.67) | 2.64 (4.32) | 1.63 (3.04)

8. Secondary Outcome: Double-Blind Period: Number of New T2 Lesions
Description: Inflammatory disease activity was assessed by MRI measurement of the number of new T2 lesions.
Time Frame: At the end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 66 | 82 | 36 | 38
lesions | 4.58 (8.36) | 3.55 (6.76) | 4.47 (6.23) | 2.42 (3.45)

9. Secondary Outcome: Double-Blind Period: Volume of T2 Lesions
Description: Volume of T2 lesion was assessed by magnetic MRI.
Time Frame: At the end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 66 | 82 | 36 | 38
cubic millimeters (mm^3) | 16930 (12816) | 17015 (15298) | 17436 (16808) | 15816 (14274)

10. Secondary Outcome: Double-Blind Period: Number of New Hypointense T1 Lesion on Enhanced T1 Scans
Description: Inflammatory disease activity was assessed by MRI measurement of the number of new hypointense T1 lesions.
Time Frame: At the end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 66 | 82 | 36 | 38
lesions | 1.23 (2.69) | 0.70 (2.01) | 1.11 (2.11) | 1.24 (2.67)

11. Secondary Outcome: Double-Blind Period: Kurtzke's Expanded Disability Status Scale (EDSS) Score
Description: EDSS (developed by John F. Kurtzke) is a scale for assessing disability in 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel and bladder, cerebral, and other functions). Each functional system score and an overall score ranges from 0 to 10, where 0 = Normal; 1-1.5 = No disability, but some abnormal neurological signs; 2-2.5 = Minimal disability; 3-4.5 = Moderate disability, affecting daily activities, but can still walk; 5-8 = More severe disability, impairing daily activities and requiring assistance with walking; 8.5-9.5 = Very severe disability, restricting to bed; 10 = Death due to MS. A lower score indicated less disability.
Time Frame: At the end of active double-blind phase or termination/early termination visit (up to Week 36)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind: Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg | Double-Blind: Placebo/Laquinimod 0.3 mg | Double-Blind: Placebo/Laquinimod 0.6 mg
Number analyzed (Participants) | 78 | 92 | 39 | 43
units on a scale | 2.53 (1.60) | 2.44 (1.21) | 2.51 (1.40) | 2.27 (1.35)

ADVERSE EVENTS:
Time Frame: Double-Blind (DB) Extension Period (Week 0 to Week 36):defined for DB treatment as start and end dates of events provided in clinical study database. Open-Label (OL) Extension Period (Month 0/termination of DB extension phase [completion of full 36 weeks] until termination [as long as Sponsor continued development of laquinimod 0.6 mg for RRMS] or early discontinuation [up to approximately 10.5 years]):defined for OL treatment as start and end dates of events provided in clinical study database.
Description: AEs that occurred after the DB end date and before OL start date are reported only once in the DB phase. AEs that occurred after the DB end date for participants who did not switch to the OL treatment are reported only once in the DB phase.
Groups:
- Double-Blind: Laquinimod 0.3 mg/Placebo to Laquinimod 0.3 mg: Participants who were receiving either laquinimod 0.3 mg or placebo matched to laquinimod 0.3 mg tablet once daily orally in double-blind core study, received laquinimod 0.3 mg tablet once daily orally in double-blind extension period of this study for up to Week 36.
- Double-Blind: Laquinimod 0.6 mg/Placebo to Laquinimod 0.6 mg: Participants who were receiving laquinimod 0.6 mg (2 tablets of 0.3 mg each) or placebo matched to laquinimod 0.6 mg (2 tablets of placebo) once daily orally in double-blind core study, received laquinimod 0.6 mg once daily orally in double-blind extension period of this study for up to Week 36.
Arm/Group | Double-Blind: Laquinimod 0.3 mg/Placebo to Laquinimod 0.3 mg | Double-Blind: Laquinimod 0.6 mg/Placebo to Laquinimod 0.6 mg | Open Label: Laquinimod 0.6 mg | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/138 | 2/113 | 0/96
Serious Adverse Events (participants affected / at risk) | 6/119 | 6/138 | 30/113 | 19/96
Other Adverse Events (participants affected / at risk) | 68/119 | 74/138 | 95/113 | 82/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind: Laquinimod 0.3 mg/Placebo to Laquinimod 0.3 mg (N=119) | Double-Blind: Laquinimod 0.6 mg/Placebo to Laquinimod 0.6 mg (N=138) | Open Label: Laquinimod 0.6 mg (N=113) | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg (N=96)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Borrelia test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular evaluation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical conisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine dilation and curettage (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subacute endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind: Laquinimod 0.3 mg/Placebo to Laquinimod 0.3 mg (N=119) | Double-Blind: Laquinimod 0.6 mg/Placebo to Laquinimod 0.6 mg (N=138) | Open Label: Laquinimod 0.6 mg (N=113) | Open-Label: Laquinimod 0.3 mg/Laquinimod 0.6 mg (N=96)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 7 (8) | 8 (13)
Tachycardia (Cardiac disorders) | 3 (3) | 6 (6) | 4 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 11 (13) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 5 (6) | 7 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 6 (6) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 3 (5) | 4 (5) | 8 (10)
Nausea (Gastrointestinal disorders) | 2 (5) | 2 (2) | 2 (2) | 5 (6)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (3) | 3 (4) | 5 (5)
Asthenia (General disorders) | 1 (1) | 2 (2) | 5 (8) | 6 (8)
Fatigue (General disorders) | 3 (3) | 4 (5) | 12 (15) | 2 (2)
Pyrexia (General disorders) | 1 (6) | 4 (4) | 6 (15) | 5 (5)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (6)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 10 (13) | 11 (14)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 8 (21) | 6 (6)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 8 (9) | 8 (9)
Nasopharyngitis (Infections and infestations) | 18 (25) | 23 (30) | 38 (96) | 39 (80)
Oral herpes (Infections and infestations) | 3 (3) | 2 (2) | 7 (15) | 7 (9)
Pharyngitis (Infections and infestations) | 5 (8) | 3 (3) | 12 (18) | 10 (21)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 10 (15) | 10 (15)
Rhinitis (Infections and infestations) | 2 (2) | 4 (4) | 7 (8) | 11 (14)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 6 (6) | 8 (15)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 3 (3) | 12 (22) | 14 (33)
Urinary tract infection (Infections and infestations) | 6 (8) | 3 (6) | 9 (11) | 8 (15)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 9 (9) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 6 (8) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 6 (8) | 1 (1)
Blood fibrinogen increased (Investigations) | 3 (3) | 6 (7) | 7 (7) | 5 (5)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2) | 8 (10) | 5 (6)
Haematocrit decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 5 (7)
Neutrophil count increased (Investigations) | 3 (3) | 1 (1) | 6 (6) | 2 (2)
White blood cell count increased (Investigations) | 3 (3) | 3 (3) | 6 (6) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (5) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 17 (22) | 10 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 12 (15) | 31 (54) | 22 (32)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 7 (9) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6) | 5 (6) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 16 (19) | 16 (20) | 17 (23) | 21 (29)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (7)
Depression (Psychiatric disorders) | 2 (2) | 1 (2) | 11 (16) | 9 (10)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (6) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 4 (6) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 5 (5) | 7 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 6 (9) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 7 (9) | 4 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5) | 5 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
Sponsor terminated RRMS studies as sufficient long term clinical data was collected for the study drug in the relevant dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT00745615/Prot_SAP_000.pdf